CLINICAL TRIAL: NCT03760068
Title: A Randomized, Multicenter, Open-Label, Parallel-Group Clinical Study Comparing the Safety and Efficacy of MYL-1601D With NovoLog® in Type 1 Diabetes Mellitus Patients
Brief Title: Mylan Insulin Aspart Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Mylan GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYL-1601D-3001
Record Dates: First submitted 2018-11-21; First posted 2018-11-30 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MYL-1601D Product (100 U/mL) (Active Comparator)
  Interventions: Drug: MYL-1601D Product
- FlexPen NovoLog® (100 U/mL) (Active Comparator)
  Interventions: Drug: FlexPen NovoLog®

INTERVENTIONS:
Drug: MYL-1601D Product — (100 U/mL)
  Arms: MYL-1601D Product (100 U/mL)
Drug: FlexPen NovoLog® — (100 U/mL)
  Arms: FlexPen NovoLog® (100 U/mL)

SUMMARY:
The aim of this phase III trial is to demonstrate the equivalence in the safety and efficacy profile between MYL-1601D and NovoLog® in patients with T1DM.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized, parallel-group phase 3 study in subjects with T1DM comparing the safety and efficacy of MYL-1601D with NovoLog®.

After up to 3-week screening period, all subjects will be titrated on NovoLog® during a 4-week run-in period, and will be shifted from their current basal insulin to study insulin Lantus®. After run-in period, subjects will be randomized; one group will receive MYL-1601D, while the other group will receive NovoLog® for 24 weeks. A follow-up visit, via telephone call, will be scheduled 4 weeks after last dose of MYL-1601D.

ELIGIBILITY:
Inclusion criteria

1. Written and signed informed consent.
2. Clinical diagnosis of type 1 diabetes mellitus for at least 6 months prior to screening.
3. Subject is able and willing to comply with the requirements of the study protocol.

Exclusion Criteria

1. History or presence of a medical condition or disease that in the Investigator's opinion would place the subject at an unacceptable risk from study participation.
2. History of hypersensitivity to any of the active or inactive ingredients of the insulin/insulin analogue preparations used in the study, OR history of significant allergic drug reactions.
3. Any clinically significant abnormality in electrocardiogram or safety laboratory tests.
4. Any elective surgery requiring hospitalization planned during the study period.
5. History of a significant medical condition, such as unstable angina, myocardial infarction, stroke or transient ischemic attack in the 6 months before screening.
6. Subjects with major depressive illness in the last 3 years.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-12-28 (Actual); Study Completion 2020-01-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (158):
- United States (158):
  - Endocrinology Associates Montgomery, Montgomery, Alabama
  - Phoenician Centers for Research, Phoenix, Arizona
  - Precision Trials, Phoenix, Arizona
  - Medical Investigations Inc., Little Rock, Arkansas
  - John Muir Physician Network, Concord, California
  - Valley Research, Fresno, California
  - Marin Endocrine Care & Research, Inc., Greenbrae, California
  - Diabetes/Lipid Management and Research Center, Huntington Beach, California
  - Diabetes And Endocrine Associates, La Mesa, California
  - Long Beach Center For Clinical Research, Long Beach, California
  - Office of Richard S. Cherlin, M.D, Los Gatos, California
  - The Rose Salter Medical Research Foundation, Newport Beach, California
  - Providence Clinical Research, North Hollywood, California
  - California Medical Research Associates Inc, Northridge, California
  - Pacific Reserach Partners, Oakland, California
  - Palmtree Clinical Research, Inc., Palm Springs, California
  - Western Univ of Health Science, Pomona, California
  - Mills-Peninsula Health Services Diabetes Research Institute, San Mateo, California
  - NorCal Endocrinology and Internal Medicine, San Ramon, California
  - Sansum Diabetes Research Institute, Santa Barbara, California
  - Coastal Biomedical Research, Inc., Santa Monica, California
  - The Metabolic Institute Of America (Mioa Inc), Tarzana, California
  - Diabetes Research Center, Tustin, California
  - Dr.Ronald H. Chochinov MD,Office Of, Ventura, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Creekside Endocrine Associates, PC, Denver, Colorado
  - New West Physicians, Golden, Colorado
  - Paradigm Research, Wheat Ridge, Colorado
  - Meridien Research, Bradenton, Florida
  - Hi Tech and Global Research, LLC, Coral Gables, Florida
  - Moonshine Research Center, Inc., Doral, Florida
  - Northeast Research Institute, Fleming Island, Florida
  - Eastern Research, Inc., Hialeah, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Care Research Center, Inc, Kendall, Florida
  - Meridien Research, Lakeland, Florida
  - Central Florida Endocrine & Diabetes Consultants, Maitland, Florida
  - Meridien Research, Maitland, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - Quality Professional Healthcare, Miami, Florida
  - Life Spring Research Foundation, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - DL Research Solutions Inc, Miami, Florida
  - Baptist Diabetes Associates, Pa, Miami, Florida
  - Medi Clear Medical & Research Center, Inc, Miami, Florida
  - Phoenix Medical Research LLC, Miami, Florida
  - Dr. De Armas Research Center, LLC, Miami, Florida
  - P & S Research, LLC, Miami, Florida
  - Inpatient Research Clinic, Miami Lakes, Florida
  - Clinical Neurosciecne Solutions, Inc. dba CNS Healthcare, Orlando, Florida
  - Omega Research Maitland, LLC, Orlando, Florida
  - Ribo Research, LLC dba Peninsula Research, Inc, Ormond Beach, Florida
  - Suncoast Clinical Research Inc., Palm Harbor, Florida
  - Hanson Clinical Research Center, Port Charlotte, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridien Research, Spring Hill, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Asclepes Research Centers, Weeki Wachee, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - IACT Health, Columbus, Georgia
  - Physicians Research Associates, LLC, Lawrenceville, Georgia
  - The Jones Center for Diabetes and Endrocrine Wellness, Macon, Georgia
  - In-Quest Medical Research, LLC, Peachtree Corners, Georgia
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Rocky Mountain Diabetes And Osteoporosis Center, Idaho Falls, Idaho
  - Advanced Clinical Research, Meridian, Idaho
  - Northwest Endo Diabets Res.LLC, Arlington Heights, Illinois
  - Midwest Endocrinology, Crystal Lake, Illinois
  - NorthShore University Health System, Skokie, Illinois
  - American Research, LLC, Jeffersonville, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Iowa Diabetes and Endocrinology Research Center (IDERC), West Des Moines, Iowa
  - Overland Park Surgical Specialties, LLC d/b/a College Park Family Care Center Physicians Group, Overland Park, Kansas
  - Cotton O'Neil Clinical Research Ctr, Topeka, Kansas
  - Veterans Affairs Medical Center, Lexington, Kentucky
  - Kentucky Diabetes And Endocrinology Center, Lexington, Kentucky
  - Crescent City Clinical Research Center, LLC, Metairie, Louisiana
  - Model Clinical Research, Baltimore, Maryland
  - Boston University School Of Medicine, Boston, Massachusetts
  - MassResearch, Waltham, Massachusetts
  - Elite Clinical Research, Flint, Michigan
  - Professional Clinical Research, Traverse City, Michigan
  - Diabetes & Endocrinology Specialists, Inc., Chesterfield, Missouri
  - Jefferson City Medical Group (Jcmg) - Jcmg Medical Building, Jefferson City, Missouri
  - Mercy Research, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Billings Clinic Research Center, Billings, Montana
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Glacier View Research Institute - Endocrinology, Kalispell, Montana
  - Diabetes & Endocrine Associates, PC Research Center, Omaha, Nebraska
  - Alegent Health Research Center, Omaha, Nebraska
  - Palm Research Center, Inc., Las Vegas, Nevada
  - Northern Nevada Endocrinology, Reno, Nevada
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - Albany Medical College, Albany, New York
  - NY Scientific, Brooklyn, New York
  - Northwell Health, Great Neck, New York
  - Scott Research,Inc, Laurelton, New York
  - Winthrop-University Hospital, Clinical Trials Center, Mineola, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Endocrine Associates of West Village, New York, New York
  - Manhattan Medical Research Practice, New York, New York
  - Dr. Jonas Leibowitz MD, Office Of, Yonkers, New York
  - Mountain Diabetes, Asheville, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Physician's East, PA, Greenville, North Carolina
  - Carteret Medical Group, Morehead City, North Carolina
  - Lucas Research, Inc., Morehead City, North Carolina
  - Medication Management, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Diabetes & Endocrinology Associates of Stark County Inc, Canton, Ohio
  - Sterling Research Group, Ltd, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Intend Clinical Research, Norman, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Endocrinology Service Northwest LLC - Bend; Advanced Specialty Care (ASC) - Bend Office, Bend, Oregon
  - Care Access Research, Warwick, Warwick, Rhode Island
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - Carolina Health Specialist, Myrtle Beach, South Carolina
  - Meridian Clinical Research, Dakota Dunes, South Dakota
  - Holston Medical Group, Bristol, Tennessee
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - WR Clinsearch, LLC, Chattanooga, Tennessee
  - Omega Research Nashville, LLC, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Amarillo Medical Specialists, Amarillo, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Baylor Research Institute, Dallas, Texas
  - UT Southwestern Medical Center Division of Endocrinology, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Academy of Diabetes Thyroid and Endocrine, El Paso, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Victorium Clinical Research, Houston, Texas
  - Juno Research, LLC, Houston, Texas
  - Endocrine IPS, PLLC, Houston, Texas
  - Clinova Clinical Trials, Houston, Texas
  - Biopharma Informatic, LLC, Houston, Texas
  - Dr.Amir Ali Hassan, MD Off of, Houston, Texas
  - North Hills Medical Research, Inc., North Richland Hills, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Science Advancing Medicine (Sam) Clinical Research, San Antonio, Texas
  - Victorium Clinical Research, San Antonio, Texas
  - Northeast Clinical Research, LLC, Schertz, Texas
  - Consano Clinical Research, Shavano Park, Texas
  - DM Clinical Research, Tomball, Texas
  - Bay Area Metabolic Health, Webster, Texas
  - Wasatch Clinical Research,LLC, Salt Lake City, Utah
  - Dr.David Gorson Md, Office Of, Bennington, Vermont
  - Manassas Clinical Research Center, Manassas, Virginia
  - Dr. Larry D. Stonesifer,MD,Office Of, Federal Way, Washington
  - Multicare Health System Research Institute, Spokane, Washington
  - The Vancouver Clinic, Inc. PS, Vancouver, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blevins TC, Raiter Y, Sun B, Donnelly C, Shapiro R, Chullikana A, Rao A, Vashishta L, Ranganna G, Barve A. Immunogenicity, Efficacy, and Safety of Biosimilar Insulin Aspart (MYL-1601D) Compared with Originator Insulin Aspart (Novolog(R)) in Patients with Type 1 Diabetes After 24 Weeks: A Randomized Open-Label Study. BioDrugs. 2022 Nov;36(6):761-772. doi: 10.1007/s40259-022-00554-6. Epub 2022 Sep 17. PMID 36114990

RESULTS

PARTICIPANT FLOW:
Groups:
- MYL-1601D Product (100 U/mL): MYL-1601D (100 U/mL) taken at mealtime. Product provided in a prefilled disposable pen with a 3-mL cartridge.
  Subjects also received during the treatment period once-daily Lantus SoloSTAR (insulin glargine injection, 100 U/mL), manufactured by Sanofi-Aventis.
- FlexPen NovoLog® (100 U/mL): FlexPen NovoLog®: (100 U/mL) taken at mealtime. Product provided in a prefilled disposable pen with a 3-mL cartridge.
  Subjects also received during the treatment period once-daily Lantus SoloSTAR (insulin glargine injection, 100 U/mL), manufactured by Sanofi-Aventis.
Period: Overall Study
Arm/Group | MYL-1601D Product (100 U/mL) | FlexPen NovoLog® (100 U/mL)
Started | 238 | 240
Completed | 224 | 217
Not Completed | 14 | 23
Not completed — Withdrawal by Subject | 7 | 8
Not completed — Adverse Event | 1 | 2
Not completed — Administrative Decision by Sponsor | 0 | 2
Not completed — Physician Decision | 1 | 2
Not completed — Lost to Follow-up | 4 | 9
Not completed — Subject Moved Out of State | 1 | 0

BASELINE CHARACTERISTICS:
Population: Type 1 Diabetes Patients
Groups:
- FlexPen NovoLog® (100 U/mL): FlexPen NovoLog® (100 U/mL) taken at mealtime. Product provided in a prefilled disposable pen with a 3-mL cartridge.
  Subjects also received during the treatment period once-daily Lantus SoloSTAR (insulin glargine injection, 100 U/mL), manufactured by Sanofi-Aventis.
- Total: Total of all reporting groups
Arm/Group | MYL-1601D Product (100 U/mL) | FlexPen NovoLog® (100 U/mL) | Total
Number analyzed (Participants) | 238 | 240 | 478
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 238 | 240 | 478
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 108 | 217
  Male | 129 | 132 | 261
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 9 | 15
  Native Hawaiian or Other Pacific Islander | 3 | 2 | 5
  Black or African American | 15 | 11 | 26
  White | 210 | 210 | 420
  More than one race | 3 | 8 | 11
  Unknown or Not Reported | 0 | 0 | 0
Screening Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.56 (4.221) | 27.00 (4.191) | 27.28 (4.211)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Emergent Antibody Response (TEAR)
Description: The number of subjects who were TEAR positive.
  TEAR is defined as either one of the following:
  1. Subjects who are Anti-Drug Antibody (ADA) negative at baseline and become positive at any timepoint post baseline
  2. Subjects who are ADA positive at baseline and demonstrate 4-fold increase in titer values at any timepoint post baseline visit.
Time Frame: Baseline to week 24
Population: Type 1 Diabetes Patients
Measure: Count of Participants; unit: Participants
Groups:
- MYL-1601D Product (100 U/mL): MYL-1601D Product: (100 U/mL) taken at mealtime. Product provided in a prefilled disposable pen with a 3-mL cartridge.
  Subjects also received during the treatment period once-daily Lantus SoloSTAR (insulin glargine injection, 100 U/mL), manufactured by Sanofi-Aventis.
Arm/Group | MYL-1601D Product (100 U/mL) | FlexPen NovoLog® (100 U/mL)
Number analyzed (Participants) | 238 | 240
Participants | 59 | 67

2. Secondary Outcome: Change in HbA1c From Baseline
Description: Mean (SD) change from baseline HbA1c at Week 24.
Time Frame: Baseline to week 24
Population: Type 1 Diabetes Patients
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | MYL-1601D Product (100 U/mL) | FlexPen NovoLog® (100 U/mL)
Number analyzed (Participants) | 238 | 240
percentage of change | 0.10 (0.735) | 0.04 (0.723)

3. Secondary Outcome: Change in Fasting Plasma Glucose From Baseline
Description: Mean (SD) change from baseline plasma glucose at Week 24.
Time Frame: Baseline to week 24
Population: Type 1 Diabetes Patients
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | MYL-1601D Product (100 U/mL) | FlexPen NovoLog® (100 U/mL)
Number analyzed (Participants) | 238 | 240
mmol/L | 0.400 (5.8162) | 0.599 (5.1553)

4. Secondary Outcome: Change in Prandial Insulin Dose From Baseline
Description: Mean (SD) change from baseline daily mealtime insulin dose at Week 24.
Time Frame: Baseline to week 24
Population: Type 1 Diabetes Patients
Measure: Mean (Standard Deviation); unit: U/kg)
Arm/Group | MYL-1601D Product (100 U/mL) | FlexPen NovoLog® (100 U/mL)
Number analyzed (Participants) | 238 | 240
U/kg) | 0.0079 (0.14608) | -0.0008 (0.09731)

5. Secondary Outcome: Change in Basal Insulin Dose From Baseline
Description: Mean (SD) change from baseline total daily insulin dose at Week 24.
Time Frame: Baseline to week 24
Population: Type 1 Diabetes Patients
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | MYL-1601D Product (100 U/mL) | FlexPen NovoLog® (100 U/mL)
Number analyzed (Participants) | 238 | 240
U/kg | 0.0053 (0.06459) | 0.0001 (0.05152)

6. Secondary Outcome: Change in Total Daily Insulin Dose From Baseline
Description: Mean (SD) change from baseline total daily insulin dose at Week 24
Time Frame: Baseline to week 24
Population: Type 1 Diabetes Patients
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | MYL-1601D Product (100 U/mL) | FlexPen NovoLog® (100 U/mL)
Number analyzed (Participants) | 238 | 240
U/kg | 0.0178 (0.15888) | 0.0024 (0.10649)

7. Secondary Outcome: Change in 7-point Self-monitored Blood Glucose (SMBG) Profile From Baseline
Description: Mean (SD) change in 7-point SMBG profile from baseline to Week 24
Time Frame: Baseline to week 24
Population: Type 1 Diabetes Patients
Measure: Mean (Standard Deviation); unit: mmol/L)
Arm/Group | MYL-1601D Product (100 U/mL) | FlexPen NovoLog® (100 U/mL)
Number analyzed (Participants) | 238 | 240
mmol/L) | 0.1180 (2.09287) | 0.0999 (1.86471)

ADVERSE EVENTS:
Time Frame: Adverse Event (AE)s or Serious Adverse Event (SAE)s were collected from the time the subject signed the informed consent form through the completion of the follow-up visit or 14 days after last dose of study medication.
Arm/Group | MYL-1601D Product (100 U/mL) | FlexPen NovoLog® (100 U/mL)
All-Cause Mortality (participants affected / at risk) | 0/238 | 1/240
Serious Adverse Events (participants affected / at risk) | 22/238 | 15/240
Other Adverse Events (participants affected / at risk) | 92/238 | 99/240
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MYL-1601D Product (100 U/mL) (N=238) | FlexPen NovoLog® (100 U/mL) (N=240)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Colititis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Incision Site Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Perineal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 15 (18) | 10 (12)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hypoglycemic Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Victim of Homicide (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MYL-1601D Product (100 U/mL) (N=238) | FlexPen NovoLog® (100 U/mL) (N=240)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 2 (3)
Nausea (Gastrointestinal disorders) | 4 (4) | 2 (2)
Food Poisoning (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Influenza Like Illness (General disorders) | 0 (0) | 3 (3)
Nasopharyngitis (Infections and infestations) | 14 (15) | 15 (19)
Upper Respiratory Tract Infection (Infections and infestations) | 11 (16) | 14 (16)
Urinary Tract Infection (Infections and infestations) | 9 (10) | 9 (11)
Sinusitis (Infections and infestations) | 1 (1) | 8 (10)
Influenza (Infections and infestations) | 0 (0) | 4 (4)
Gastroenteritis (Infections and infestations) | 0 (0) | 3 (3)
Weight Increased (Investigations) | 3 (3) | 4 (4)
Blood Pressure Increased (Investigations) | 3 (5) | 3 (3)
Glycosylated Hemoglobin Increased (Investigations) | 3 (3) | 1 (1)
Crystal Urine Present (Investigations) | 0 (0) | 3 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5) | 5 (6)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Headache (Nervous system disorders) | 9 (13) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Orophayngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-10-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT03760068/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT03760068/SAP_001.pdf